CLINICAL TRIAL: NCT07389044
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics, And Preliminary Efficacy of Single and Multiple Ascending Doses of IB-001 in Healthy Participants and Participants With Chronic Hepatitis B
Brief Title: A Study on IB-001 Dose Response and Tolerability in Healthy Adults and Those With Chronic Hepatitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IntegerBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IB001-001
Record Dates: First submitted 2026-01-16; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B Virus Infection
Keywords: First in Human; Single Ascending Dose; Multiple Ascending Dose; Hepatitis B virus; HBV; Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: IB-001 (Experimental): Participants receive IB-001, administered subcutaneously according to the assigned cohort schedule. In Part A (SAD), participants receive a single ascending dose. In Part B (MAD), participants receive once-weekly dosing for 4 weeks.
  Interventions: Drug: IB-001
- Arm 2: Placebo (Placebo Comparator): Participants receiving placebo subcutaneously, following the same dosing schedule as the active arm (single dose in SAD; once-weekly for 4 weeks in MAD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IB-001 — Subcutaneous (SC) injectable formulation; single ascending dose in HVs (Part A) and multiple ascending weekly doses for 4 weeks in CHB participants (Part B). Exact dose levels recommended by SRC review.
  Arms: Arm 1: IB-001
Drug: Placebo — Subcutaneous (SC) injection; no active ingredients.
  Arms: Arm 2: Placebo

SUMMARY:
This study will examine the safety and tolerability of single and multiple doses of IB-001, and will be conducted in two parts:

Part A: SAD study in approximately 60 Healthy Volunteer (HV). Part B: MAD study in approximately 30 adult participants living with Chronic Hepatitis B (CHB).

DETAILED DESCRIPTION:
This is a first-in-human, double-blind, randomized, placebo-controlled Phase 1 study of IB-001 administered subcutaneously to evaluate safety, tolerability, PK/PD, and preliminary antiviral activity.

The study is comprised of two parts:

Part A: Single Ascending Dose (SAD) in Healthy Volunteers Up to 60 healthy adult participants in up to six cohorts (n=10 per cohort; 8 active:2 placebo). Participants will receive a single sub-cutaneous dose of investigational product followed by a 28-day post treatment follow-up. .

Part B: Multiple Ascending Dose (MAD) in Treatment-Naïve or Currently-Not-Treated Adults with Chronic Hepatitis B (CHB) Up to 30 adult participants (3 cohorts; n=10 per cohort; 8 active:2 placebo). Once-weekly sub-cutaneous dosing over 4 weeks with 6-week post-treatment follow-up. Dose recommendations in both Part A and Part B will be made by the Safety Review Committee (SRC) based on review of emerging safety data.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Male or female aged 18 to 70 years.
3. Females must not be of childbearing potential OR those who are of childbearing potential must be non-pregnant and non-lactating and willing to use a highly effective method of contraception.

   Males whose partners are of childbearing potential must either be surgically sterile or willing to use a highly effective acceptable method of contraception.
4. Non-tattooed, clear injection site suitable for SC injection and monitoring in the opinion of the Investigator.

Exclusion Criteria:

Healthy participants must not meet any of the following criteria at Screening or upon admission to the site (on Day -1).

1. Major surgery requiring general anesthesia within 12 weeks prior to Screening or is expected to have surgery requiring general anesthesia during the course of the study.
2. History of severe allergic or anaphylactic reactions, or sensitivity to the IP or its constituents.
3. Blood donation or blood loss of ≥ 1 unit (450 mL) of whole blood within 4 weeks before Screening or plasma donations within 7 days prior to dosing on Study Day 1.
4. Any underlying medical condition (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrinological, tumor, pulmonary, immune, mental, or cardiovascular and cerebrovascular diseases).
5. History of malignancy, except for non-melanoma skin cancer, excised more than 1 year prior to Screening or cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening.
6. Current hepatitis A virus (HAV) infection, hepatitis B virus (HBV) infection , hepatitis C virus (HCV) infection , or hepatitis E virus (HEV) infection .Positive test for HIV-1 or HIV-2 antibodies.
7. Any other active infection requiring systemic antiviral or antimicrobial therapy that will not be completed within 2 weeks of first dosing.
8. Clinically significant 12-lead ECG abnormalities on Screening ECG.
9. History of cardiac arrhythmias.
10. Physical examination findings at Screening that are considered clinically significant by the Investigator and likely to adversely impact study conduct and/or interpretation.
11. Clinically significant abnormal vital signs
12. Laboratory examination abnormalities considered clinically significant by the Investigator at Screening.
13. Use of any prescribed or over-the-counter medications (including vitamins or herbal remedies) within 2 weeks of first dosing or within 5 times the elimination half-life of the medication prior to first dosing.
14. Any suspicion or history of drug and/or alcohol abuse within the last year.
15. Pregnant, planning to become pregnant during the course of the study, or currently breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-04 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs). | Through Day 29 (Part A), through Day 64 (Part B).
  Treatment-Emergent Adverse Events (TEAEs) are adverse events that first appear or worsen in severity during the course of the clinical study, regardless of whether they are related to the investigational product (IP) or not. TEAEs will be coded using MedDRA and summarized by SOC, PT, severity, and relationship to IP. Treatment-related AEs (possibly/probably/definitely related) will also be summarized separately. A by-participant AE listing will be provided
Part A and Part B: Number of Participants with Adverse Events (AEs) by Severity | Through Day 29 (Part A), through Day 64 (Part B)
  An AE is any unfavorable medical occurrence in a study participant administered an investigational product. The AE does not necessarily have a causal relationship with the treatment. All AEs will be graded for severity according to NCI-CTCAE classification. If an appropriate AE term is not found in NCI-CTCAE, the AE will be graded as follows: Grade 1 (mild); Grade 2 (Moderate); Grade 3 (Severe); Grade 4 (Severe) and Grade 5 (Death).
Part A and Part B: Number of Participants with Adverse Events (AEs) of Special Interest (AESIs) | Through Day 29 (Part A), through Day 64 (Part B)
  AEs of special interest include Cytokine Release Syndrome (CRS), Injection Site Reactions (ISRs) and Unexplained Liver Biochemistry Elevations. Reported AESIs will be graded according to NCI-CTCAE classification. If an appropriate AE term is not found in NCI-CTCAE, the AESI will be graded as follows: Grade 1 (mild); Grade 2 (Moderate); Grade 3 (Severe); Grade 4 (Severe) and Grade 5 (Death).
Part A and Part B: Number of Participants with Clinically Significant Changes in Laboratory Parameters | Through Day 15 (Part A), through Day 64 (Part B)
  Assessment Method - Number of participants with clinical laboratory abnormalities (serum chemistry, hematology, and coagulation) will be reported.
Part A and Part B: Number of Participants with Clinically Significant Changes in Vital Signs. | Through Day 15 (Part A), through Day 64 (Part B)
  Number of participants with vital signs abnormalities will be reported. Vital signs include body temperature, pulse rate, respiratory rate, and blood pressure.
Part A and Part B: Number of Patients with Clinically Significant Changes in Cardiac Parameters. | Through Day 15 (Part A), through Day 64 (Part B)
  Number of participants with electrocardiogram (ECG) abnormalities will be reported.

SECONDARY OUTCOMES:
Part A and Part B: Number of Patients with Clinically Significant Anti-Drug Antibodies (ADAs). | Through Day 29 (Part A), through Day 64 (Part B)
  All immunogenicity data (ADA) are to be analyzed using the Immunogenicity Analysis Population. ADA incidence and titer levels over time will be summarized by dose.
Part B: Changes from Baseline in HBsAg levels over time. | Through Day 64 (Part B)
  Blood samples will be analyzed for HBsAg levels to establish baseline and determine eligibility; subsequent blood samples will be collected at protocol-specified timepoints to measure HBsAg changes over time.
Part B: Change from Baseline in Anti-HBs Antibody Titers over time. | Through Day 64
  Blood samples will be collected at baseline and at protocol-specified timepoints to measure anti-HBs antibody titer changes over time.
Part B: Reduction from Baseline in HBV DNA levels over time. | Through Day 64
  Blood samples will be collected at baseline and at protocol-specified timepoints to measure HBV DNA changes over time.
Part A and Part B: PK Parameter - Maximum Observed Serum Concentration (Cmax) of IB-001 | Through Day 29 (Part A), through Day 64 (Part B)
  The Cmax is the maximum observed concentration of IB-001 in serum following single or multiple ascending dose administration. Blood samples will be collected at baseline and at protocol-specified timepoints.
Part A and Part B: PK Parameter - Area under the Serum Concentration Time Curve (AUC) of IB-001. | Through Day 29 (Part A), through Day 64 (Part B)
  AUC is the area under the concentration time curve of IB-001 in serum following single or multiple ascending dose administration. Blood samples will be collected at baseline and at protocol-specified timepoints.
Part A and Part B: PK Parameter - Time to Observed Maximum Serum Concentration (Tmax) of IB-001. | Through Day 29 (Part A), through Day 64 (Part B)
  Tmax is the time it takes to reach maximum concentration of IB-001 in serum following single or multiple ascending dose administration. Blood samples will be collected at baseline and at protocol-specified timepoints.
Part A and Part B: PK Parameter - Terminal Half Life (T1/2) of IB-001. | Through Day 29 (Part A), through Day 64 (Part B)
  T1/2 will be measured following single and multiple doses of IB-001. Blood samples will be collected at baseline and at protocol-specified timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Gane, MBChB, MD, FRACP, MNZ, Principal Investigator — New Zealand Clinical Research
Locations (1):
- New Zealand Clinical Research, Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No